CLINICAL TRIAL: NCT07122141
Title: Validity and Reliability of the 6-Minute Pegboard and Ring Test in Interstitial Lung Disease
Status: Active, not recruiting | Type: Observational
Sponsor: Marmara University (Other)
Responsible Party: Principal Investigator, Anıl Gökçen, Physiotherapist, Marmara University
Other Study IDs: Upperextremity_ILD
Record Dates: First submitted 2025-08-07; First posted 2025-08-14 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Interstitial Lung Diseases (ILD)
Keywords: 6-minute pegboard and ring test; upper extremity; validity; reliability; Interstitial lung diseases (ILD)
MeSH Terms: conditions — Lung Diseases, Interstitial

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this study is to investigate the validity and reliability of the 6 Minutes Pegboard and Ring Test (6PBRT) in patients with Interstitial Lung Disease (ILD).

DETAILED DESCRIPTION:
Our study was conducted in the Chest Diseases Clinic of Süreyyapaşa Chest Diseases and Thoracic Surgery Training and Research Hospital. Our study was approved by the Marmara University Faculty of Health Sciences Non-Interventional Clinical Research Ethics Committee and was conducted in accordance with the Declaration of Helsinki. Signed informed consent was obtained from the participants.

ELIGIBILITY:
Inclusion Criteria:

* who were diagnosed with ILD according to the ATS/ERS/JRS/ALAT guidelines,
* were over 18 years of age,
* had not changed their treatment for the last 3 months,
* had a stable clinical status for the last 3 months.

Exclusion Criteria:

* Neurological comorbidity,
* Orthopedic comorbidity that impairs upper extremity function,
* Kyphoscoliosis and/or severe postural abnormalities,
* Uncontrolled cardiac problems,
* Uncontrolled diagnosis of Diabetes Mellitus,
* Ischemic heart disease,
* Newly diagnosed history of cancer,
* Diagnosis of obstructive pulmonary disease,
* Cognitive impairments such as Alzheimer's or dementia,
* Use of immunosuppressive medications (excluding corticosteroids),
* History of recent surgery,
* Refusal to answer questions,
* Refusal to participate voluntarily.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Chest Diseases Clinic of Süreyyapaşa Chest Diseases and Thoracic Surgery Training and Research Hospital
Sampling Method: Probability Sample
Enrollment: 27 (Estimated)
Dates: Start 2025-04-25 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
6 Minutes Pegboard and Ring Test (6PBRT) | Day 1
  The 6-Minute Pegboard and Ring Test (6PBRT) is designed to assess upper extremity functional capacity using unsupported arm movements. The setup includes four horizontally aligned bars: two at shoulder height and two positioned 20 cm above. Participants, seated with back support, sequentially transfer rings between the bars for six minutes, and the total number of rings moved serves as the performance score.
6 Minutes Walking Tests (6MWT) | Day 1
  Total distance walked (in meters) during the 6MWT will be recorded. Higher distance reflects improved functional capacity.
Unsupported Upper-Limb Exercise Test (UULEX) | Day 1
  Patients will be instructed to lift five bars consecutively and rhythmically until the onset of fatigue. The bars will have incremental weights of 200 g, 500 g, 1 kg, and 2 kg, respectively. The duration of the activity will be recorded to assess the patients' endurance levels.

SECONDARY OUTCOMES:
1 Minute Sit to Stand Test (1MSTST) | Day 1
  The 1-Minute Sit-to-Stand Test (1MSTST) is a simple, inexpensive, and practical assessment used to evaluate functional capacity in a small space. During the test, participants are asked to repeatedly sit down and stand up from a fixed chair as quickly as possible for one minute, without using their arms for support.
Spirometric measurements (Forced vital capacity - FVC) | Day 1
  It is used to assess respiratory function and is measured using a spirometer. Forced Vital Capacity (FVC) refers to the maximum volume of air that can be forcefully exhaled from the lungs after a full inhalation. This value can be expressed in liters or as a percentage.
Spirometric measurements (First second forced expiratory volume - FEV1) | Day 1
  It is employed to assess respiratory functions and is measured using a spirometer. Forced Expiratory Volume in the first second (FEV₁) represents the volume of air that can be forcefully exhaled within the first second of a maximal exhalation. This parameter can be expressed either in liters or as a percentage.
Spirometric measurements (FEV1/FVC ratio) | Day 1
  It is employed to assess respiratory function and is measured with a spirometer. The value is obtained by dividing FEV₁ by FVC, and the result is expressed as a percentage.
Carbon monoxide diffusion capacity | Day 1
  Carbon monoxide diffusion capacity (DLCO) is the measurement of the passage of carbon monoxide gas in inspired air into the lung capillary blood. Diffusion test is performed in the pulmonary function test laboratory.
Gender-Age-Physiology (GAP) Index | Day 1
  The Gender-Age-Physiology (GAP) index is a multidimensional assessment index developed and validated to predict mortality in ILD. The ILD-GAP index is divided into stages 0-1, 2-3, 4-5, and >5, which predict the risk of death in the 1st, 2nd, and 3rd years. The GAP index will be calculated based on gender (0-1 points), age (0-2 points), %FVC (0-2 points), and %DLCO (0-3 points). It is classified into Stage I (0-3 points), Stage II (4-5 points), and Stage III (6-8 points), with prognosis worsening as it progresses from Stage I to Stage III.
Modified Medical Research Council Dyspnea Score | Day 1
  The Modified Medical Research Council (mMRC) Dyspnea Scale assesses the sensation of breathlessness as perceived by the individual. The severity of dyspnea is scored on a scale ranging from 0 to 4, where 0 indicates no perception of dyspnea and 4 represents severe breathlessness.
Handgrip Strength | Day 1
  A manual hydraulic dynamometer will be used for the hand grip strength test, taking into account the recommendations of the American Association of Occupational Therapists (AAOT). During the test, measurements will be taken while the patient is seated with back support, shoulder in adduction and neutral position, elbow at 90° flexion, and forearm in neutral position.
Fatigue severity scale | Day 1
  he fatigue levels of individuals will be evaluated using the Fatigue Severity Scale. This scale comprises nine items rated on a 7-point Likert scale, reflecting the individual's perception of fatigue, which may indicate the need for medical intervention. The total score is 63. Higher scores indicate more severe fatigue.
London Chest Daily Activities of Living Scale | Day 1
  The feeling of breathlessness experienced during daily living activities was assessed using the London Chest Daily Activities of Living Scale (LCADL). The scale consists of a total of 15 items divided into four sections: personal care (4 items), housework (6 items), physical activity (2 items), and leisure activities (3 items). Each item is scored on a scale of 0-5. The total score for the scale is 75. A high score indicates an increased perception of shortness of breath during daily living activities.
Saint George Quality of life questionnaire | Day 1
  The St. George's Respiratory Questionnaire is designed to assess health-related quality of life in individuals with respiratory conditions. It provides four separate scores: Symptoms, Activity, Impacts, and an overall Total score. The scale ranges from 0 to 100, where 0 represents no impairment in quality of life and 100 indicates the most severe impairment.

CONTACTS AND LOCATIONS:
Overall Officials: Anıl Gökçen, Phsiotheraphist, Principal Investigator
Locations (1):
- Süreyyapaşa Chest Diseases and Thoracic Surgery Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No